CLINICAL TRIAL: NCT02102802
Title: Exploring Mechanisms of Action of ±3,4-methylenedioxymethamphetamine (MDMA)- Assisted Psychotherapy for Posttraumatic Stress Disorder (PTSD)
Brief Title: Exploring Mechanisms of Action in MDMA-assisted Psychotherapy for PTSD
Status: Completed | Type: Observational
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: MP8-S1
Record Dates: First submitted 2014-03-27; First posted 2014-04-03 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; MDMA; Brain activity; fMRI; Heart rate variability; Physiological correlate
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Therapeutics

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MDMA-assisted therapy: Participants undergoing MDMA-assisted therapy in the main study, MP-8 (NCT#01211405)
  Interventions: Drug: Midomafetamine; Behavioral: Therapy

INTERVENTIONS:
Drug: Midomafetamine — 125, 75, or 30 mg midomafetamine HCl followed 1.5 to 2 hours later by a supplemental dose of midomafetamine HCl half the initial dose
  Other Names: 3,4-methylenedioxymethamphetamine; MDMA
Behavioral: Therapy — Manualized therapy

SUMMARY:
The goal of this observational sub-study is to provide information on how MDMA-assisted therapy affects the brain and body of people with chronic PTSD.

The main question it aims to answer is: Is PTSD symptom reduction associated with changes in heart rate variability and brain activity?

Participants from the MP-8 study will be invited to enroll in this sub-study where they will undergo an fMRI brain scan and other measurements of body function.

DETAILED DESCRIPTION:
This exploratory sub-study will identify psychotherapeutic processes occurring during MDMA- assisted psychotherapy in people with chronic PTSD and assess the feasibility of exploring physiological correlates of clinical outcomes in subjects enrolled in the ongoing clinical trial of MDMA-assisted psychotherapy, NCT #: NCT01211405. The sub-study will be conducted in collaboration with researchers at the Medical University of South Carolina (MUSC), Smith College and the New School for Social Research.

To support the clinical outcomes measured by CAPS from the MP-8 study, the sponsor is interested in correlations of outcomes with treatment-related changes in potential biological markers of PTSD, measured by heart rate variability (HRV) and fMRI. Brain activity while listening to neutral and personalized trauma-related scripts will take place at baseline and after experimental MDMA-assisted psychotherapy with low, medium, or full dose MDMA. The fMRI scan will be followed by a Diffusion Tensor Imaging (DTI) scan. After each scanning session, pulse measurements will be extracted as a digital data file from which HRV will be calculated. FMRI scans and HRV measurements will occur at baseline for participants in all conditions, one month after the second experimental session and again after a final experimental session for participants in the low or medium dose condition, and two months after the final experimental session for participants in the full dose condition.

Participants will complete the Self-Compassion Scale, a self-report measure of self-compassion at Baseline and after the final MDMA-assisted psychotherapy session. Psychotherapeutic processes will be assessed via observing psychotherapy and sorting a set of 100 therapy-related items as a means of describing the interactions. Trained coders will observe at least one pre-drug psychotherapy session, one experimental (drug-assisted psychotherapy) session and one post-drug psychotherapy session.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the parent study, "A Randomized, Triple-Blind, Phase 2 Pilot Study Comparing 3 Different Doses of MDMA in Conjunction with Manualized Psychotherapy in 24 Veterans, Firefighters, and Police Officers with Chronic, Treatment-Resistant Posttraumatic Stress Disorder (PTSD)." NCT #: NCT01211405

Exclusion Criteria:

* Mass brain lesion
* Have metal in their skulls,
* Having brain or heart pacemakers
* History of major head trauma
* Have past or present panic or extreme discomfort with being in small enclosed spaces (claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants enrolled in the parent study, MP-8
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08-03 (Actual); Study Completion 2015-08-03 (Actual)

PRIMARY OUTCOMES:
Change in brain activity measured via fMRI while listening to trauma scripts | Baseline, two months after final experimental session
  Brain activity measured via functional magnetic resonance imaging (fMRI) after listening to trauma-related scripts.

SECONDARY OUTCOMES:
Change in heart rate variability in response to trauma script | Baseline, one month post-drug
  Assessment of Heart rate variability (HRV) in response to trauma-related scripts; a potential physiological correlate of response to treatment for PTSD
Change in Self Compassion Scale Score | Baseline, one month post-drug
  Self-report measure of self-compassion
Change in heart rate variability in response to trauma script | Baseline, two months post final drug administration
  Assessment of Heart rate variability (HRV) in response to trauma-related scripts; a potential physiological correlate of response to treatment for PTSD
Change in Self Compassion Scale Score | Baseline, two months post final drug administration
  Self-report measure of self-compassion
Change in brain activity measured via fMRI while listening to trauma scripts | Baseline, one month post-drug
  Brain activity measured via functional magnetic resonance imaging (fMRI) after listening to trauma-related scripts

OTHER OUTCOMES:
Psychotherapy Process Q-set (PSQ) | 3 - 7 weeks post enrollment
  System of coding psychotherapeutic processes in observed psychotherapy (pre-drug)
Psychotherapy Process Q-set (PSQ) | 8 - 16 weeks post-enrollment
  System of coding psychotherapeutic processes in observed psychotherapy (drug-assisted psychotherapy session)
Psychotherapy Process Q-set (PSQ) | 17-27 weeks post-enrollment
  System of coding psychotherapeutic processes in observed psychotherapy (end of treatment after final experimental session)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Mithoefer, MD, Principal Investigator — Private Practice
Locations (1):
- Offices of Michael Mithoefer, Mt. Pleasant, South Carolina, United States

REFERENCES:
- [Derived] Singleton SP, Wang JB, Mithoefer M, Hanlon C, George MS, Mithoefer A, Mithoefer O, Coker AR, Yazar-Klosinski B, Emerson A, Doblin R, Kuceyeski A. Altered brain activity and functional connectivity after MDMA-assisted therapy for post-traumatic stress disorder. Front Psychiatry. 2023 Jan 12;13:947622. doi: 10.3389/fpsyt.2022.947622. eCollection 2022. PMID 36713926

DOCUMENTS (1):
  • Informed Consent Form (2013-12-03): https://cdn.clinicaltrials.gov/large-docs/02/NCT02102802/ICF_000.pdf